CLINICAL TRIAL: NCT06888375
Title: Humidification Practices During Non-Invasive Ventilation in Hospitalized Patients: A Multinational Survey
Brief Title: Humidification Practices During Hospitalized Patients on Non-Invasive Ventilation
Acronym: NIV
Status: Completed | Type: Observational
Sponsor: Dr. Ram Manohar Lohia Hospital (Other Government)
Collaborators: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government); Hospital General Universitario Morales Meseguer (Other)
Responsible Party: Principal Investigator, Sanjay Singhal, sanjay, Dr. Ram Manohar Lohia Hospital
Other Study IDs: IEC No. 244/24; RC1779 (Other: RESEARCH CELL, Dr. Ram Manohar Lohia Institute of Medical Sciences, Lucknow (India))
Record Dates: First submitted 2025-03-15; First posted 2025-03-21 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-04

CONDITIONS: Acute Respiratory Disease; Non Invasive Ventilation (NIV)
Keywords: NIV; Humidification; Acute respiratory failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physicians dealing with adult patients with acute respiratory failure: to assess the practice pattern of humidification use among physicians during NIV in hospitalized adult patients

SUMMARY:
To date, the practice pattern of humidification during Non-Invasive Ventilation (NIV) is unknown. This study aims to assess the practice pattern of physicians regarding humidification use in hospitalized adult patients on NIV. This study will recognize the gaps between current practice and available evidence.

Primary Objective:

(a) Prevalence of Humidification use and their types

Secondary Objective:

1. Reasons for not using humidification
2. Reasons for choosing a specific humidification device

DETAILED DESCRIPTION:
Non-invasive ventilation (NIV) provides respiratory support through a mask compared to invasive mechanical ventilation (IMV) using an endotracheal or tracheostomy tube. NIV has become a standard of care in managing acute respiratory failure, especially in acute exacerbation of chronic obstructive pulmonary disease, acute cardiogenic pulmonary edema, immunocompromised patients, and weaning from IMV. Over the past few decades, its use has increased drastically in these patients, reducing the need for IMV, morbidity, and mortality. However, various studies have reported NIV failure in 20-50% of patients owing to poor tolerance. Non-humidified inspired gases used in NIV and IMV are very dry, and their humidification can prevent their harmful effect on the respiratory system. Heat and Humidification in IMV is the standard of care worldwide, but no consensus or guidelines regarding its use during NIV. Although the upper airways are not bypassed in NIV, physiological air conditioning could be insufficient due to circuit leaks, high respiratory drive, a high fraction of inspired oxygen (FiO2), type of mask, mouth breathing, and use of dry air with ICU ventilators. Inadequate humidification in hospitalized patients with acute respiratory failure using NIV can lead to difficult intubation after NIV failure, life-threatening airway obstruction due to thick secretions, and increased airway reactivity. Based on various physiological and clinical studies, AARC clinical practice guidelines suggested humidification in patients with NIV. To date, the practice pattern of humidification during NIV is unknown.

This study aims to assess the practice pattern of physicians regarding humidification use during NIV in hospitalized adult patients. This study will recognize the gaps between current practice and available evidence.

Objective:

Primary Objective:

(a) Humidification utilization rate and their types

Secondary Objective:

1. Reasons for not using humidification
2. Reasons for choosing a specific humidification device

Methodology:

1. Study design: This is a cross-sectional web-based survey among physicians who are dealing with NIV. Participation will be on an invitation basis and purely voluntary after informed consent.
2. Inclusion criteria: Physicians dealing with adult patients with acute respiratory failure
3. Exclusion criteria: Physicians who refuse to give consent
4. Study Duration: six months
5. Study setting: A pre-designed survey link will be sent to all members of the various respiratory and critical care societies. Each physician who consented to participate will receive a web-based questionnaire. Physicians who did not respond to the first email within eight weeks will receive reminders.
6. Sample Size: As per a survey by Crimi C et al.14, humidification was used in more than 50% of clinical scenarios using NIV. We calculate our sample size by using the formula N= t.p.q/ε2 where N is equal to the required sample size, t is similar to the confidence level at 95% (standard value of 1.96), p is equal to estimated prevalence (humidification use), q is equal to 1-prevalence, ε is similar to allottable error. Using the above formula in the prevalence of 50%, our sample size is 384. We will exclude responses like not using NIV, incomplete data (>10%), and working in the same unit. We added 20% to compensate for this, so our final sample size would be 462.
7. Data Analysis: Data will be collected, compiled, and analyzed using IBM-SPSS-29 software. Descriptive statistics (mean, median, and proportions) will be used to report survey questionnaire responses. The Kruskal-Walli's test will be used for non-parametric data to evaluate the variability depending on the physician's primary specialty and hospital setting.
8. Consent: The invited email will have details of the study purpose and a participant information sheet. An email will also contain a Google Form link with instructions that implied consent will be considered if they agree to participate and submit their response.

ELIGIBILITY:
Inclusion Criteria:

* Physicians dealing with adult patients with acute respiratory failure with NIV

Exclusion Criteria:

* Physicians who refuse to give consent or not using NIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: web-based survey among physicians dealing with NIV in adult patients with acute respiratory failure
Sampling Method: Probability Sample
Enrollment: 534 (Actual)
Dates: Start 2025-04-19 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Humidification utilization rate and their types | six months
  Humidification utilization rate will be calculated by a total number of respondents using humidification during NIV in patients with acute respiratory failure divided by a total number of respondents involved in managing patients of acute respiratory failure on NIV. Details will also be collected regarding the type of humidification type (Heated humidifier or Heat Moisture Exchange (HME)).

SECONDARY OUTCOMES:
Reasons for not using humidification | six months
  Details about the reasons for not using humidification during NIV use will also will be collected.
Reasons for choosing a specific humidification device | six months
  Depending upon their preference of humidification devices (Heated humidifier or HME), details will also be collected for the reasons about their preference.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio M Esquinas, MD, PhD, FCCP, FNIV, Study Chair — School of Non-invasive Mechanical Ventilation Hospital Morales Meseguer, Murcia, Spain
Locations (2):
- India (2):
  - Dr Sanjay Singhal, Lucknow, Uttar Pradesh
  - Dr. Ram Manohar Lohia Institute of Medical Sciences, Lucknow, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in non-invasive ventilation. Shared Data will be coded, with no PHI included. Approval of the request and execution of all applicable agreements are prerequisites for sharing the data with the requesting party.
Supporting Information: Study Protocol, SAP
Time Frame: six months after publication
Access Criteria: Data requests can be submitted starting six months after publication and up to 24 months. Extensions will be considered on a case-to-case basis.